CLINICAL TRIAL: NCT02783742
Title: Teaching Provider Communication Via Coaching to Reduce Burnout
Brief Title: Provider-Patient Communication Coaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00072714
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Provider Burnout; Communication
Keywords: provider-patient communication; coaching; feedback; burnout
MeSH Terms: conditions — Communication; Burnout, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Providers in this arm will receive a communication coaching intervention immediately post-randomization.
  Interventions: Behavioral: Communication coaching
- Waitlist Control (Other): Providers assigned to this arm will be offered the option of receiving the communication coaching intervention after follow up data collection is complete.
  Interventions: Behavioral: Communication coaching

INTERVENTIONS:
Behavioral: Communication coaching — Study coaches will conduct tailored individual sessions with participating providers to teach and improve communication techniques. Coaches will then shadow or audio-record patient encounters and deliver feedback to providers on their communication during these encounters.

SUMMARY:
To examine the effect of a coaching intervention on provider burnout and communication

DETAILED DESCRIPTION:
The investigator will recruit providers at Duke University and randomly assign them to receive (1) a communication coaching intervention or (2) a waitlist intervention. The investigator will survey all providers at Baseline and Follow Up. Providers randomized to the intervention arm will attend face-to-face meetings with study coaches, and have some of their encounters with patients shadowed by a coach or audio recorded. Providers will obtain verbal consent from patients to participate in the study (i.e. have their encounter shadowed or audio recorded). Providers will then be provided feedback by coaches on their communication during these encounters. Providers randomized to the waitlist intervention arm will be offered the option of receiving this intervention after they complete the follow up survey.

ELIGIBILITY:
Inclusion Criteria:

* Providers and patients at Duke University Medical Center

Exclusion Criteria:

* Younger than 18
* non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Change in provider burnout, as measured by questionnaire | baseline and follow up, approximately 2 months

SECONDARY OUTCOMES:
change in comfort addressing emotion, as measured by questionnaire | baseline and follow up, approximately 2 months
change in self-rated efficiency, as measured by questionnaire | baseline and follow up, approximately 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pollak KI, Gao X, Beliveau J, Griffith B, Kennedy D, Casarett D. Pilot Study to Improve Goals of Care Conversations Among Hospitalists. J Pain Symptom Manage. 2019 Nov;58(5):864-870. doi: 10.1016/j.jpainsymman.2019.06.007. Epub 2019 Aug 16. PMID 31422103